CLINICAL TRIAL: NCT06997705
Title: Strengthening HPV Vaccination and Adolescent Health Research Program (SHARP) in Ivory Coast
Brief Title: Integrated HPV Vaccination and Adolescent Health in Ivory Coast
Acronym: SHARP-CI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 30593
Record Dates: First submitted 2025-03-31; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Integrated Care; HPV Vaccination; Adolescent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized VMS (Experimental): The intervention arm will receive an optimized integrated adolescent health service package, including HPV vaccination - this will included newly introduced modalities/modifications in school, health facility, and community settings.
  Interventions: Behavioral: Optimized VMS
- VMS (comparison) (No Intervention): The comparison arm will receive routine health services for adolescents with no programmatic changes. Routine health services delivered to school and university adolescent and youth are part of a program called the Systematic Medical Visit (VMS).

INTERVENTIONS:
Behavioral: Optimized VMS — Building on the Systematic Medical Visits (VMS) the Optimized VMS, optimizes these services for in-school and out-of-school adolescents by expanding availability of VMS services through community and facility platforms and building capacity of health workers to provide integrated services. Also the intervention will involve demand generation activities such as community sensitization.
  Other Names: SHARP-intervention in Cote d'Ivoire
  Arms: Optimized VMS

SUMMARY:
Background: Cervical cancer is a serious global public health problem, particularly in sub-Saharan Africa, where it is the leading cause of cancer in women, with around 70,722 new cases each year. Vaccination against human papillomavirus (HPV) prevents cervical cancer and is usually given to children around 9 to 15 years of age. HPV vaccination has been incorporated into many countries' Expanded Programs on Immunization, but often faces optimization and uptake challenges. SHARP is an implementation research initiative in Tanzania, Nigeria, and Côte d'Ivoire that is looking at the potential of combining HPV vaccination with with adolescent primary care/preventive health services - how this might work and its effect on the uptake of the HPV vaccine and other services.

Objective: To describe the feasibility, acceptability, effectiveness and sustainability of a locally-designed integrated adolescent health service package, including HPV vaccination in Cote d'Ivoire. Specifically, this study aims to optimize existing primary health care approaches, making service delivery not only more convenient but also more effective in addressing the specific needs of adolescents-both in school and out of school-across schools, communities, and health facilities.

Methods: This is a quasi-experimental research study using the difference-in-difference method between an intervention group and a comparison group over time. It will use mixed methods drawing on quantitative surveys, qualitative interviews, service time motion assessment, and administrative data. The study will be conducted in two regions, each with an intervention and comparison district. The optimized adolescent integrated health intervention will be implemented in the intervention districts with routine service provision in comparison areas. Monthly administrative service coverage data and baseline and endline surveys will be conducted in up to 3502 households with 1626 parents/caregivers and 1626 adolescents will assess effectiveness by looking at changes in service uptake and coverage, as well in knowledge, attitudes, and practices towards HPV vaccination and integrated services. At endline, up to 132 in-depth interviews will be conducted with program managers, health officials, service providers, school authorities, community influencers and leaders, and adolescents and parents/caregivers will assess feasibility, acceptability and sustainability.

ELIGIBILITY:
Inclusion Criteria for adolescents:

* Age: 9 to 15;
* Residence in the study regions;
* Parental or guardian permission is required;
* Provides assent and agrees to participate in the study.

Inclusion criteria for Parents/caregivers:

* Be the parent or legal guardian of an adolescent aged 9 to 15 years;
* Residence in the study regions;
* Provides informed consent and agrees to participate in the study.

Exclusion Criteria:

* People who have time constraints;
* those who do not speak French or the prominent dialects in study regions;
* those unable to participate because ill, intoxicated or appearing psychologically impaired;
* those residing outside study health regions;
* those who do not provide consent/assent to participate.

Ages: 9 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3384 (Estimated)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number/proportion of adolescent girls vaccinated for HPV | Baseline (before intervention start) and at endline (up to 8 months after intervention); regularly collected information from registers will be collected by study team members on a montly basis during interverntion
  This is an effectiveness measure that captures the HPV coverage among adolescent girls residing in the study areas.
Number/proportion of adolescent girls intending to get HPV vaccine | Baseline (before intervention start) and at endline (6 months after intervention)
  This measure, captured through the survey, aggregates those who have received HPV vaccination in the past 6 months as well as those who express an intention to get vaccinated in the next 6 months.

SECONDARY OUTCOMES:
Number/proportion of participants with HPV knowledge | Baseline (before intervention start) and at endline (6 months after intervention)
  This measure will be captured through a survey by several knowledge related items, including an adapted composite measure (standardized scale: Human Papillomavirus Knowledge Questionnaire (PHV-KQ)).
Number/proportion of participants with positive attitudes towards integrated services | Baseline (before intervention start) and at endline (6 months after intervention)
  This outcome reflects several indicators related to attitudes related to accessing integrated adolescent health services, including HPV vaccination assessed through several items on a questionnaire (not a validated scale).

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Charurat, MBA, MHS, Principal Investigator — Jhpiego
Locations (1):
- École Nationale Supérieure de Statistique et d'Économie Appliquée (ENSEA), Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: No